CLINICAL TRIAL: NCT03176186
Title: XePOHCAS - Xenon by Inhalation for Post Out of Hospital Cardiac Arrest Syndrome
Brief Title: Xenon for Neuroprotection During Post-Cardiac Arrest Syndrome in Comatose Survivors of an Out of Hospital Cardiac Arrest
Acronym: XePOHCAS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Invero Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XePOHCAS Ph III
Record Dates: First submitted 2016-12-05; First posted 2017-06-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Post-Cardiac Arrest Syndrome
Keywords: ischemic-reperfusion injury; out of hospital cardiac arrest
MeSH Terms: conditions — Post-Cardiac Arrest Syndrome; Out-of-Hospital Cardiac Arrest | interventions — Xenon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- TH/TTM (No Intervention): Protocol-directed standard of care (including TH/TTM) dictated by the 2015 guidelines for Post-Cardiac Arrest Care from the American Heart Association and the European Resuscitation Council. Mechanical Ventilation delivered by individual site-sanctioned ventilator.
- TH/TTM plus Xenon (Active Comparator): 50% xenon gas in addition to standard of care, including therapeutic hypothermia/targeted temperature management (TH/TTM).
  Interventions: Combination Product: Xenon

INTERVENTIONS:
Combination Product: Xenon — 50% xenon by inhalation, delivered by customized xenon delivery system, that includes a ventilator, for the 24h period of TH/TTM. The inhalation therapy is provided in combination with protocol-directed Post-Cardiac Arrest Care dictated by the 2015 guidelines from the American Heart Association and the European Resuscitation Council.
  Other Names: XENEX
  Arms: TH/TTM plus Xenon

SUMMARY:
XePOHCAS: Prospective, randomized, multicenter interventional trial in adult subjects with out-of-hospital cardiac arrest comparing treatment with standard-of-care post-cardiac arrest intensive care (which is targeted temperature management [TTM]) to xenon by inhalation plus standard-of-care post-cardiac arrest intensive care (including TTM).

DETAILED DESCRIPTION:
XePOHCAS:

Primary Objective:

To evaluate whether there is a difference in functional outcome with xenon 50% and oxygen during targeted temperature management (TTM) compared with similar oxygen content in air during TTM in comatose subjects with sustained restoration of spontaneous circulation (ROSC) within 30 minutes after out-of-hospital cardiac arrest (OHCA).

Secondary Objective:

To evaluate whether there is a difference in survival with xenon 50% and oxygen during targeted temperature management (TTM) compared with similar oxygen content in air during TTM in comatose subjects with sustained restoration of spontaneous circulation (ROSC) within 30 minutes after out-of-hospital cardiac arrest (OHCA).

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years but less than or equal to 80 years
2. Presumed cardiac cause of arrest
3. Sustained (>20 minutes) spontaneous circulation upon arrival in the emergency department
4. No response to verbal commands on arrival to emergency department and prior to randomization (Glasgow Coma Scale score of <8)
5. Attending decision that patient is eligible for TTM

Exclusion Criteria:

1. Written do not attempt resuscitation reported to providers before randomization
2. Traumatic etiology of arrest, defined as concomitant blunt, penetrating, or burn-related injury, or uncontrolled bleeding or exsanguination
3. Suspected or known stroke or intracranial hemorrhage
4. Unwitnessed cardiac arrest
5. No-flow (cardiac arrest to initiation of cardiopulmonary resuscitation/defibrillation) time of >10 minutes
6. Sustained restoration of spontaneous circulation (ROSC) greater than 30- minutes post-arrest
7. Interval from arrival at the emergency department to randomization for intervention of >4 hours.
8. Hypothermia (<30°C core temperature)
9. Bed-bound prior to cardiac arrest
10. Unconsciousness before cardiac arrest (cerebral trauma, spontaneous cerebral hemorrhage, intoxication etc.)
11. Coagulopathy
12. Systolic arterial pressure <80 mmHg or mean arterial pressure <60 mmHg lasting more than 30 minutes after ROSC
13. Known pregnancy
14. Have received an investigational drug, device, or biologic product within 30-days
15. Known terminal phase of chronic illness
16. Hypoxemia (SaO2 <85%) for >15 minutes after ROSC
17. Inability to maintain SaO2 >90% on an FiO2 of 50%
18. Having any other clinically significant laboratory abnormality, medical condition (such as intrinsic liver disease or severe chronic obstructive pulmonary disease), or social circumstance that, in the investigator's opinion, makes it inappropriate for the patient to participate in this clinical trial
19. Logistically impossible to provide intervention
20. Have any condition that would impact the evaluation of modified Rankin Scale (mRS)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1436 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
functional outcome: degree of functional independence measured using a modified Rankin Scale (mRS) | 30 days after the cardiac arrest
  The degree of functional independence will be measured using a modified Rankin Scale (mRS)

SECONDARY OUTCOMES:
survival: number of survivors | 30 days after the cardiac arrest
  The number of survivors will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Stuerzebecher, M.D., Study Director — CMO Invero Pharma
Locations (10):
- United States (8):
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - University Nebraska Medical Center, Omaha, Nebraska
  - University at Buffalo, Buffalo, New York
  - Wexner Medical Center, Ohio State University, Columbus, Ohio
  - Baptist Memorial Hospital, Baptist Clinical Research Institute, Memphis, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - University Hospital, Rigshospitalet, Blegdamsvej 9, Copenhagen

IPD SHARING:
Plan to Share IPD: Yes
Authorized representatives of the SITE OF STUDY CONDUCT or other associated health care providers as authorized.

REFERENCES:
- [Background] Laitio R, Hynninen M, Arola O, Virtanen S, Parkkola R, Saunavaara J, Roine RO, Gronlund J, Ylikoski E, Wennervirta J, Backlund M, Silvasti P, Nukarinen E, Tiainen M, Saraste A, Pietila M, Airaksinen J, Valanne L, Martola J, Silvennoinen H, Scheinin H, Harjola VP, Niiranen J, Korpi K, Varpula M, Inkinen O, Olkkola KT, Maze M, Vahlberg T, Laitio T. Effect of Inhaled Xenon on Cerebral White Matter Damage in Comatose Survivors of Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2016 Mar 15;315(11):1120-8. doi: 10.1001/jama.2016.1933. PMID 26978207
- [Derived] Magliocca A, Fries M. Inhaled gases as novel neuroprotective therapies in the postcardiac arrest period. Curr Opin Crit Care. 2021 Jun 1;27(3):255-260. doi: 10.1097/MCC.0000000000000820. PMID 33769417
- See also: Phase 2 RCT that forms the basis for this clinical trial — http://jamanetwork.com/journals/jama/fullarticle/2503174